CLINICAL TRIAL: NCT04250636
Title: An Open Label, Single Arm Study of the Safety, Pharmacokinetics and Antiretroviral Activity of the Combination of 3BNC117-LS and 10-1074-LS in Viremic HIV-infected Individuals.
Brief Title: 3BNC117-LS and 10-1074-LS in Viremic HIV-infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Weill Medical College of Cornell University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCA-0994; 1U01AI145921 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: 3BNC117-LS; 10-1074-LS; Broadly Neutralizing Antibody
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): HIV-infected individuals, off ART, and with plasma HIV-1 RNA levels between 500 and 100,000 copies/ml by standard assays. Study participants will receive a single intravenous infusion of 3BNC117-LS and a single infusion of 10-1074-LS. The antibodies will be administered sequentially and dosed at 30 mg/kg.
  Interventions: Drug: 3BNC117-LS; Drug: 10-1074-LS

INTERVENTIONS:
Drug: 3BNC117-LS — Intravenous infusion of 3BNC117-LS at 30mg/kg
  Other Names: Monoclonal Antibody
Drug: 10-1074-LS — Intravenous infusion of 10-1074-LS at 30mg/kg
  Other Names: Monoclonal Antibody

SUMMARY:
The proposed study is a phase 1, open label, single arm study to evaluate the safety, pharmacokinetics and antiviral activity of single intravenous infusions of 3BNC117-LS and 10-1074-LS, each monoclonal antibody (mAb) dosed at 30 mg/kg in viremic human immunodeficiency virus (HIV)-infected individuals.

DETAILED DESCRIPTION:
The proposed study is a phase 1, open label, single arm study to evaluate the safety, pharmacokinetics and antiviral activity of single intravenous infusions of 3BNC117-LS and 10-1074-LS in viremic HIV-infected individuals.

Ten eligible participants will be enrolled sequentially in the study and will receive each mAb, dosed at 30 mg/kg intravenously and in sequence on study day 0. Following mAb administration, study participants will return for safety assessments on days 1 and 3, and weeks 1, 2, 3 and 4 following dosing, then bi-weekly or monthly until the end of study follow up. All participants will be followed for 24 weeks after 3BNC117-LS and 10-1074-LS administration.

Safety assessments will be performed at multiple time points following 3BNC117-LS and 10-1074-LS infusions. Serum samples for pharmacokinetic (PK) measurements will be collected before and at the end each mAb infusion administration and at multiple subsequent time points during study follow up. Samples will also be collected for measurement of HIV-1 plasma RNA levels before 3BNC117-LS and 10-1074-LS infusions (screen and day 0) and at every follow up visit. T cell subsets will also be monitored during study follow up. Assessments will also include measurement of anti-drug antibody responses and sequencing of plasma envelope before infusions and after viral rebound (first time point after viremia nadir is reached and viral load (VL) is > 1,000 copies/ml).

Participants will be advised and encouraged to start antiretroviral therapy (ART) within 4 weeks of receiving 3BNC117-LS and 10-1074-LS infusions or sooner if: VL fails to decrease by > 0.5 log10 copies/ml within 2 weeks of antibody infusions, VL increases > 0.5 log10 copies/ml between weekly measurements or significant T-cell decline (confirmed CD4+ T cells < 200 cells/μl) is noted.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, >18 years of age.
2. Confirmed HIV-1 infection.
3. Off ART for at least 4 weeks with a HIV-1 plasma RNA level between 500 and 100,000 copies/mL (ART-naïve or off ART due to intolerance or by choice).
4. Current CD4+ T cell count > 300 cells/μl.
5. If sexually active male or female, and participating in sexual activity that could lead to pregnancy or transmission of HIV, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom) from 10 days prior to and six months after 3BNC117-LS and 10-1074-LS administration.

Exclusion Criteria:

1. Have a history of AIDS-defining illness within 3 years prior to enrollment.
2. History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
3. Any clinically significant acute or chronic medical condition (such as autoimmune diseases), other than HIV infection, that in the opinion of the investigator would preclude participation.
4. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
5. Laboratory abnormalities in the parameters listed below:

   * Absolute neutrophil count ≤ 1,000 cells/μl;
   * Hemoglobin ≤ 10 gm/dL;
   * Platelet count ≤ 100,000 cells/μl;
   * ALT ≥ 1.5 x ULN;
   * AST ≥ 1.5 x ULN;
   * Alkaline phosphatase ≥ 1.5 x ULN;
   * Total bilirubin > 1.25 x ULN;
   * eGFR < 60 mL/min/1.73m2.
6. Pregnancy or lactation.
7. Any vaccination within 14 days prior to mAb infusions, except for influenza vaccine.
8. Receipt of another investigational product currently or within the past 12 weeks, or expected concurrent participation in another study in which investigational products will be administered.
9. Receipt of any experimental HIV vaccine or anti-HIV monoclonal antibody therapy in the past.
10. History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
11. Individuals with known hypersensitivity to any constituent of the investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, Principal Investigator — The Rockefeller University
Locations (3):
- United States (3):
  - Weill Cornell Medical Center Clinical Trials Unit-CLOSED SITE, New York, New York
  - The Rockefeller University, New York, New York
  - Perelman School of Medicine University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open-label, sequential enrollment
Period: Overall Study
Arm/Group | Study Participants
Started | 6
Completed | 4
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 35.8 [26 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 and Serious Adverse Events
Description: The number of participants with treatment-related solicited and unsolicited grade 3 and serious adverse events (including confirmed laboratory abnormalities).
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Peak Concentration
Description: Peak concentration of 3BNC117-LS and 10-1074-LS when administered intravenously and in combination to viremic HIV-infected individuals.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Study Participants
Number analyzed (Participants) | 6
mcg/ml
  3BNC117-LS | 719.83 (77.62)
  10-1074-LS | 915.15 (207.18)

3. Primary Outcome: Half-life
Description: Half-life of 3BNC117-LS and 10-1074-LS when administered intravenously and in combination to viremic HIV-infected individuals.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Participants
Number analyzed (Participants) | 6
days
  3BNC117-LS | 41.63 (11.71)
  10-1074-LS | 47.62 (15.38)

4. Primary Outcome: Area Under Curve
Description: Area under curve of 3BNC117-LS and 10-1074-LS when administered intravenously and in combination to viremic HIV-infected individuals.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: (mcg x day)/mL
Arm/Group | Study Participants
Number analyzed (Participants) | 6
(mcg x day)/mL
  3BNC117-LS | 13965.98 (2922.99)
  10-1074-LS | 34539.92 (34539.92)

5. Primary Outcome: Maximum Decline in Plasma HIV-1 RNA Level
Description: Maximum decline in plasma HIV-1 RNA level after 3BNC117-LS plus 10-1074-LS intravenous infusions in viremic HIV-infected individuals through week 4 after infusions.
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: log 10 HIV-1-RNA copies/ml
Arm/Group | Study Participants
Number analyzed (Participants) | 6
log 10 HIV-1-RNA copies/ml | 1.79 [1.1 to 2.4]

6. Secondary Outcome: Anti-drug Antibodies
Description: Number of individuals with treatment-induced anti-drug antibodies against each mAb and magnitude of the response.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 6
Participants
  Anti-3BNC117-LS | 0
  Anti-10-1074-LS | 1

7. Secondary Outcome: Adverse Events
Description: The number of adverse events that occur during the study follow up period after 3BNC117-LS and 10-1074-LS administration.
Time Frame: 24 weeks
Measure: Number; unit: adverse events
Arm/Group | Study Participants
Number analyzed (Participants) | 6
adverse events | 5

8. Secondary Outcome: Laboratory Abnormalities
Description: The number of confirmed laboratory abnormalities that occur during the study follow up period after 3BNC117-LS and 10-1074-LS administration.
Time Frame: 24 weeks
Measure: Number; unit: graded laboratory abnormalities
Arm/Group | Study Participants
Number analyzed (Participants) | 6
graded laboratory abnormalities | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 weeks.
Description: Definitions are the definitions of CT.gov
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=6)
Tinea capitis (Infections and infestations) | 1 (1)
Pyrosis (Gastrointestinal disorders) | 1 (1)
Penile trauma (Injury, poisoning and procedural complications) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT04250636/Prot_SAP_000.pdf